CLINICAL TRIAL: NCT03626298
Title: Efficacy and Tolerability of Nicotinamide Plus Cream for Moderate Acne Vulgaris in Indonesia: A Multicenter Clinical Trial
Brief Title: Efficacy and Tolerability of Nicotinamide Plus Cream for Moderate Acne Vulgaris in Indonesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rumah Sakit Pusat Angkatan Darat Gatot Soebroto (Other)
Responsible Party: Principal Investigator, Dr Irma Bernadette S Sitohang, Medical Doctor, Rumah Sakit Pusat Angkatan Darat Gatot Soebroto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PapulexPaper1
Record Dates: First submitted 2018-07-17; First posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene; Niacinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adapalene and placebo (ADAP) (Placebo Comparator)
  Interventions: Drug: Adapalene; Drug: Placebos
- Adapalene, Nicotinamide, ABA, Zinc PCA (ANAZ) (Experimental)
  Interventions: Drug: Adapalene; Drug: Nicotinamide, ABA and Zinc PCA

INTERVENTIONS:
Drug: Adapalene — third-generation topical retinoid primarily used in the treatment of mild-moderate acne. It is effective against acne conditions where comedones are predominant.
Drug: Nicotinamide, ABA and Zinc PCA — combination of three non-antibiotic active ingredients of nicotinamide, anti-bacterial adhesive agent (ABA) and zinc, or abbreviated as ANAZ to be well-tolerated by patients with acne vulgaris
  Arms: Adapalene, Nicotinamide, ABA, Zinc PCA (ANAZ)
Drug: Placebos — Placebo cream. to resemble an active medication or therapy so that it functions as a control; this is to prevent the recipient(s) and/or others from knowing (with their consent) whether a treatment is active or inactive, as expectations about efficacy can influence results.
  Arms: Adapalene and placebo (ADAP)

SUMMARY:
Acne vulgaris (AV) is a chronic inflammatory disease of the pilosebaceous unit that affects seborrheic areas such as the face, back and chest. AV is characterized by blackheads, papules, pustules nodes and cysts with sequelae of hyperpigmentation and scarring. It is one of the most common skin disorders treated by dermatologists. Acne vulgaris can be found at any age, although it is more frequent in teenagers and young adults. The prevalence of AV in a population of 11 to 30 years old is approximately 80%. Due to its involvement of the face, it is considered to be a cosmetic problem, thus bearing a psychosocial burden.

ELIGIBILITY:
Inclusion Criteria:

* moderate acne vulgaris
* 12 and up to 50 years old,
* agreed to become research participants and has signed the informed consent.

Exclusion Criteria:

-

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 125 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
inflammatory and non-inflammatory acne lesion reduction number analyzed using GLMM | 6 weeks
  objective evaluation was based on photographs of participants from three angles per visit. The outcome of efficacy was measured from the percentage reduction of inflammatory and non-inflammatory lesions number and analyzed using the GLMM (General Linear mixed Model)

IPD SHARING:
Plan to Share IPD: No